CLINICAL TRIAL: NCT02693574
Title: Comparison Efficacy of 14-day Triple Therapy Between Clarithromycin and Levofloxacin on the Eradication of Helicobacter Pylori in Syrian Population
Brief Title: Comparison Efficacy of 14-day Triple Therapy: Clarithromycin vs. Levofloxacin on Eradication of H. Pylori
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Damascus Hospital (Other)
Collaborators: UNIPHARMA. Universal Pharmaceutical Industries (Unknown); Ibn Alhaytham Pharma. Industries Co (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G1
Record Dates: First submitted 2016-02-11; First posted 2016-02-26 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-01

CONDITIONS: Helicobacter Pylori Gastrointestinal Tract Infection
Keywords: Helicobacter pylori; Helicobacter Infections; Proton Pump Inhibitors
MeSH Terms: conditions — Helicobacter Infections | interventions — Clarithromycin; Esomeprazole; Amoxicillin; Levofloxacin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clarithromycin (Active Comparator): Clarithromycin 500 mg Tablets and Esomeprazole 20 mg Capsule And Amoxicillin 1000 mg,Tablets by mouth every 12 hours for 14 days
  Interventions: Drug: Clarithromycin
- Levofloxacin (Experimental): Levofloxacin 500 mg coated tablets and Esomeprazole 20 mg Capsule and Amoxicillin 1000 mg Tablets by mouth every 12 hours for 14 days
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: Clarithromycin
  Other Names: Esomeprazole; Amoxicillin
  Arms: Clarithromycin
Drug: Levofloxacin
  Other Names: Esomeprazole,Amoxicillin; Amoxicillin
  Arms: Levofloxacin

SUMMARY:
Comparison Efficacy of 14-day Triple Therapy between Clarithromycin and levofloxacin on the Eradication of Helicobacter Pylori in Syrian population

ELIGIBILITY:
Inclusion Criteria:

1-Patients are aged greater than 18 years old who have H. pylori infection diagnosed by any of following three methods: I-Positive rapid urease test (CLOtest). II-Histologic evidence of H. pylori by modified Giemsa staining. III-Positive 13C-urea breath test. without prior eradication therapy and are willing to receive therapy.

Exclusion Criteria:

1. Children and teenagers aged less than 18 years.
2. Previous eradication treatment for H. pylori.
3. Patients who took any drug, which could influence the study results such as proton pump inhibitor, H2 blocker, mucosal protective agent and antibiotics.
4. History of gastrectomy.
5. Gastric malignancy, including adenocarcinoma and lymphoma,
6. Previous allergic reaction to antibiotics (Amoxicillin, Clarithromycin, Levofloxacin) and prompt pump inhibitors (Es-omeprazole).
7. Contraindication to treatment drugs.
8. Pregnant or lactating women.
9. Severe concurrent disease.
10. Liver cirrhosis.
11. Chronic kidney disease.
12. Patients who cannot give informed consent by himself or herself.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-01-28 (Actual); Study Completion 2017-05-31 (Estimated)

PRIMARY OUTCOMES:
Eradication rate according to Intention to treat (ITT) and per-protocol (PP) analysis | 6 weeks after eradication therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Damascus Hospital, Damascus, Syria

IPD SHARING:
Plan to Share IPD: Undecided